CLINICAL TRIAL: NCT02465905
Title: Oral Immunotherapy in Cow's Milk Allergy (CMA) in Children : "Petit Lait" Study
Acronym: Petit Lait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Flore AMAT (Other)
Responsible Party: Sponsor-Investigator, Dr Flore AMAT, MD, Association Poumon et Enfance
Organization: Association Poumon et Enfance (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-A00641-42
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raw milk (Active Comparator): For raw milk immunotherapy (RMI), fixed dose of raw milk was daily administered at home, determined using tolerated threshold dose during the DBPCFC. Augmentation was made every 5 weeks in the allergy clinic.
  Interventions: Other: raw milk
- Heated milk (Active Comparator): For heated milk immunotherapy (HMI), families were asked to weekly increase the daily dose of milk at home using industrial preparations. Milk included in the preparation was less and less heated among time. Passage from heated-milk to half-heated milk and then raw milk was performed in the allergy clinic.
  Interventions: Other: Heated milk

INTERVENTIONS:
Other: raw milk
  Arms: Raw milk
Other: Heated milk
  Arms: Heated milk

SUMMARY:
Prospective study Main objective: to evaluate the efficiency and the security of two protocols of immunotherapy (raw milk versus heated milk) in a cohort of children with persistent Immunoglobulin E (IgE) mediated CMA (IgE-CMA).

Secondary objectives: to determinate if the enumeration of casein-specific IL-4- and IL-13-secreting T cells could be a valuable biomarker of successful immunotherapy.

DETAILED DESCRIPTION:
The study prospectively included children aged older than 3 years, with an IgE-CMA.

Children were part of the " Petit Lait " Study, led from June 2012 in the Allergology Department of Armand Trousseau Children's Hospital, "Assistance Publique-Hôpitaux de Paris (AP-HP)", France

1. Inclusion criteria All the children presenting with a diagnosis of IgE- CMA(defined as a history of reaction to the ingestion of cow's milk product and positive skin prick test (wheal ≥3 mm to cow's milk with no reaction to the negative control and specific IgE to casein >0.35 (kiloUnit) kU/l) and referred to one of the Allergology Department were offered to enter the study.

   Double-blind, placebo-controlled (DBPCFC) oral food challenge The DBPCFC was performed outside of episodes of exacerbation of acute illness. Children were admitted to the allergy clinic on two separate days, and food challenges were performed under the supervision of an experienced allergist. A peripheral intravenous line was inserted in each patient before starting the challenge, according to recommendations.Increasing doses of cow's milk were administered 20 min apart. Two protocols were available, one called " standard protocol " and one called "hyperallergic protocol". Type of protocol was chosen before inclusion through a multidisciplinar and collegial manner. Challenge was stopped in case of a clinical reaction compatible with an allergic reaction. Antihistamine, methylprednisolone, bronchodilator or epinephrine was administered if necessary. Cumulative dose of cow's milk tolerated defined the reactive threshold in CMA children.
2. Exclusion criteria Children who have presented an anaphylactic reaction during the previously year, who reacted with placebo during the DBPCFC or those with lacking consent or parents having difficulties to understand the protocol were excluded from the study.
3. Oral Immunotherapy Phase Children were assigned by randomization to raw milk immunotherapy or heated milk immunotherapy.
4. Prospective follow-up A monthly call was performed by a medical staff trained to allergology and families were asked on milk dose daily ingested at home and on eventual adverse side effects. A final DBPCFC using the standard protocol was planned once the daily dose attained 80 mL of raw milk.
5. Biological markers

   * Measurement of IgE and Immunoglobulin G4 (IgG4) against casein
   * Measurement of Interleukin 4 (IL4) and Interleukin 13 (IL13) secreting lymphocyts by an Enzym Link ImmunoSpot (ELISpot) assay to cow's milk protein

ELIGIBILITY:
Inclusion Criteria:

* All the children presenting with a diagnosis of IgE- CMA(defined as a history of reaction to the ingestion of cow's milk product and positive skin prick test (wheal ≥3 mm to cow's milk with no reaction to the negative control and specific IgE to casein >0.35 kU/l)

Exclusion Criteria:

* Children who have presented an anaphylactic reaction during the previously year, who reacted with placebo during the DBPCFC or those with lacking consent or parents having difficulties to understand the protocol

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome: increased tolerance to cow's milk | 12 months
  daily unit dose in milliliters of milk ingested
Clinical Outcome: occurrence of allergic reaction to cow's milk | 12 months
  Number of patients with occurrence of allergic reaction; if yes, severity of allergic reaction evaluated using: Astier score; number of use of rescue medications such as: bronchodilator, anti-histaminics, systemic corticosteroids, epinephrin

SECONDARY OUTCOMES:
Biological Outcome: kinetics of specific IgE against casein | 12 months
  changes in blood level of specific IgE against casein
Biological Outcome: kinetics of specific IgG4 against casein | 12 months
  changes in blood level of specific IgG4 against casein
Biological Outcome: kinetics of IL4 secreting lymphocytes against casein | 12 months
  ELISPOT assay
Biological Outcome: kinetics of IL13 secreting lymphocytes against casein | 12 months
  ELISPOT assay

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Allergologie, Paris, France